CLINICAL TRIAL: NCT02632786
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study of NEOD001 in Previously Treated Subjects With Light Chain (AL) Amyloidosis Who Have Persistent Cardiac Dysfunction
Brief Title: The PRONTO Study, a Global Phase 2b Study of NEOD001 in Previously Treated Subjects With Light Chain (AL) Amyloidosis
Acronym: PRONTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOD001-201
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: AL Amyloidosis
Keywords: amyloidosis; ntprobnp; NEOD001; Prothena; PRONTO; amyloid; plasma cell dyscrasia; immunotherapy
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis; Alzheimer Disease; Paraproteinemias | interventions — birtamimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NEOD001 (Experimental): Study Drug given IV every 28 days at 24mg/kg
  Interventions: Drug: NEOD001
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NEOD001 — NEOD001 is a monoclonal antibody directed at soluble and insoluble light chain aggregates
  Arms: NEOD001
Drug: Placebo — Saline Bag
  Arms: Placebo

SUMMARY:
This is a global, multicenter, Phase 2b, randomized, double-blind, placebo-controlled, two-arm, parallel-group efficacy and safety study of NEOD001 as a single agent administered intravenously in adults with AL amyloidosis who had a hematologic response to previous treatment for their amyloidosis (e.g., chemotherapy, autologous stem cell transplant [ASCT]) and have persistent cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Confirmed diagnosis of systemic AL amyloidosis
3. ≥1 prior systemic plasma cell dyscrasia therapy with at least a partial hematologic response
4. Cardiac involvement
5. NT-proBNP ≥650

Exclusion Criteria:

1. Non-AL amyloidosis
2. Meets the International Myeloma Working Group (IMWG) definition of Multiple Myeloma
3. NT-proBNP >5000
4. Received Plasma cell directed chemotherapy within 6 months
5. Received autologous stem cell transplant (ASCT) within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (19):
  - City of Hope, Duarte, California
  - Stanford Cancer Institute (SCI), Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas; MD Anderson Cancer Center, Houston, Texas
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Cancer Center - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - The University of Queensland - Princess Alexandra Hospital (PAH), Woolloongabba, Queensland
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
- Medizinische Universität Wien, Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- France (4):
  - Hôpital Dupuytren - CHU Limoges, Limoges
  - Hôpital Pitié-Salpêtrière, Paris
  - Hopitaux Lyon Sud, Pierre-Bénite
  - CHU Rennes, Service de Medecine Interne, Rennes
- Germany (4):
  - Charite-Universitatsmedizin, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitatsklinikum Hamburg-Eppendorf (UKE, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
- Greece (2):
  - Alexandra General Hospital of Athens, Athens
  - University Hospital of Patras, Pátrai
- Hadassah University Medical Center, Jerusalem, Israel
- Policlinica San Matteo, Pavia, Italy
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
- United Kingdom (3):
  - Centre for Clinical Haematology, Birmingham
  - The Royal Free London NHS Foundation Trust - The Royal Free Hospital, London
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- NEOD001 24mg/kg: NEOD001, 24 mg/kg IV every 4 weeks for 12 months
- Placebo: Placebo, 0.9% Saline IV every 4 weeks for 12 months
Period: Overall Study
Arm/Group | NEOD001 24mg/kg | Placebo
Started | 66 | 63
Informed Consent Obtained | 66 | 63
Randomized and Dosed | 66 | 63
Completed | 55 | 56
Not Completed | 11 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Death | 3 | 2
Not completed — Physician Decision | 5 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEOD001 24mg/kg | Placebo | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 29 | 70
  >=65 years | 25 | 34 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.09 (9.188) | 63.90 (8.332) | 62.98 (8.794)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 39 | 39 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 64 | 61 | 125
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 3 | 2 | 5
  Race: White | 61 | 56 | 117
  Race: Other | 1 | 3 | 4
  Race: Multiple Races Reported | 0 | 0 | 0
  Race: Not reported | 0 | 2 | 2
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiac Response and Non-Response
Description: N-terminal pro-brain natriuretic peptide (NT-proBNP ) best response (Response or Non-Response [Stable, Progression]) from baseline through 12 months of treatment. Cardiac best response, as assessed by NT-proBNP alone, is defined as the most favorable category among response (ie, decrease in NT-proBNP from baseline of >30% and >300 ng/L), stable (ie, neither response nor progression), and progression (ie, increase in NT-proBNP from baseline of >30% and >300 ng/L) across all visits after the first infusion of study drug up to and through the end of the study. Subjects are considered non-responders until a response is achieved. Non-response is defined as either stable or progression.
Time Frame: Baseline through 12 months of treatment
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | NEOD001 24mg/kg | Placebo
Number analyzed (Participants) | 66 | 63
Participants
  Response | 26 | 30
  Non-response | 40 | 33
Statistical Analysis 1: Comparison: NEOD001 24mg/kg; Test type: Superiority; p = 0.3190, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.55 to 1.21]

2. Secondary Outcome: SF-36v2 PCS Score
Description: Change in Short Form-36 (SF-36 version 2) questionnaire Physical Component Summary [PCS] Score. PCS scores are calculated based on responses to specific Short Form-36 (version 2) questions using a weight scoring method. The lower the PCS score the more disability, the higher the score the less disability. A score of 50 is the mean in the US General Population and the standard deviation is 10. Minimum is 0 and maximum value is 100.
Time Frame: Baseline to 12 months of treatment
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NEOD001 24mg/kg | Placebo
Number analyzed (Participants) | 66 | 63
score on a scale | 0.19 [-1.83 to 2.22] | 0.97 [-0.99 to 2.93]
Statistical Analysis 1: Comparison: NEOD001 24mg/kg vs Placebo; Test type: Superiority; p = 0.5563, Mixed Models Analysis; Mean Difference (Net) = -0.78, 95% CI 2-sided [-3.37 to 1.81]

3. Secondary Outcome: 6MWT Distance
Description: Change in 6 Minute Walk Test (6MWT) Distance (meters)
Time Frame: Baseline to 12 months of treatment
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- NEOD001 24 mg/kg: NEOD001, 24 mg/kg IV every 4 weeks for 12 months
Arm/Group | NEOD001 24 mg/kg | Placebo
Number analyzed (Participants) | 66 | 63
meters | 19.25 [-21.75 to 59.37] | 8.00 [-24.99 to 47.24]
Statistical Analysis 1: Comparison: NEOD001 24 mg/kg vs Placebo; Test type: Superiority; p = 0.8992, ANCOVA; Mean Difference (Net) = 5.00, 95% CI 2-sided [-11.50 to 23.00]

4. Secondary Outcome: Number of Participants With Renal Best Response and Non-Response
Description: Proteinuria and estimated Glomerular Filtration Rate (eGFR) response (Response or Non-Response [Stable, Progression]) from baseline through 12 months of treatment in subjects with renal involvement. Renal best response, as assessed by proteinuria, is defined as the most favorable category among response (ie, ≥30% decrease from baseline or <0.5 g/24 hours postbaseline result if subject does not meet criteria for progression), stable (ie, neither response nor progression), and progression (ie, ≥25% decrease in eGFR from baseline) across all visits after the first infusion of study drug up to and through the end of the study. Subjects are considered non-responders until a response is achieved. Assessments that qualify as both a response and progression are counted as progression.
  Non-response is defined as either stable or progression.
Time Frame: Baseline through 12 months of treatment
Population: Renal Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | NEOD001 24 mg/kg | Placebo
Number analyzed (Participants) | 13 | 18
Participants
  Response | 7 | 6
  Non-Response (Stable, Progression) | 6 | 12
Statistical Analysis 1: Comparison: NEOD001 24 mg/kg vs Placebo; Test type: Superiority; p = 0.3529, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.54, 95% CI 2-sided [0.60 to 3.94]

5. Secondary Outcome: NIS-LL Total Score
Description: Change in Neuropathy Impairment Score-Lower Limb (NIS-LL) Total Score in subjects with peripheral nerve involvement. NIS-LL is a scoring system graduated from 0 points to a maximum of 88 points (the absence of all motor, sensory, and reflex activity in the lower extremities). The scale is an additive of all deficits (64 potential points for muscle strength, 8 points for reflexes, and 16 points for sensory function) in the lower extremities. A score of 0 is normal and score of 88 is total impairment.
Time Frame: Baseline to 12 months of treatment
Population: Peripheral Neuropathy Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NEOD001 24 mg/kg | Placebo
Number analyzed (Participants) | 12 | 14
score on a scale | -1.2 [-3.9 to 1.6] | -0.6 [-3.0 to 1.8]
Statistical Analysis 1: Comparison: NEOD001 24 mg/kg vs Placebo; Test type: Superiority; p = 0.7570, Mixed Models Analysis; Mean Difference (Net) = -0.6, 95% CI 2-sided [-4.2 to 3.0]

6. Secondary Outcome: NT-proBNP Slope
Description: Rate of change in NT-proBNP (ng/L per infusion). Estimates of the intercept, slope, SE, and associated 95% CI for each treatment group, and the NEOD001 and placebo group difference comparisons are estimated using a general linear mixed effects model. The model fits a random intercept and slope for each subject and includes fixed effects for treatment group, time, treatment group by time interaction, IWRS stratification factors (hematologic response to first-line therapy: CR/VGPR, PR and NT-proBNP <1800 ng/L, ≥1800 ng/L), and an unstructured covariance structure to model the within-subject errors. Time is represented in months as a continuous variable and includes all scheduled time points, including baseline. The p-value is associated with the visit by treatment group interaction term.
Time Frame: Baseline through 12 months of treatment
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: ng/L per infusion
Arm/Group | NEOD001 24 mg/kg | Placebo
Number analyzed (Participants) | 66 | 63
ng/L per infusion | 9.45 [-45.66 to 64.55] | 81.41 [25.15 to 137.68]
Statistical Analysis 1: Comparison: NEOD001 24 mg/kg vs Placebo; Test type: Superiority; p = 0.0729, Mixed Models Analysis; Slope = -71.97, 95% CI 2-sided [-150.72 to 6.79]

7. Secondary Outcome: Hepatic Best Response
Description: Alkaline Phosphatase response (Response or Non-Response [Stable, Progression]) from baseline through 12 months of treatment in subjects with hepatic involvement
Time Frame: Baseline through 12 months of treatment
Population: Hepatic Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | NEOD001 24 mg/kg | Placebo
Number analyzed (Participants) | 5 | 4
Participants
  Response | 1 | 0
  Non-response | 4 | 4
Statistical Analysis 1: Comparison: NEOD001 24 mg/kg vs Placebo; Test type: Superiority; p = 0.4142, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Initiation of study drug through the last study visit or up to 30 days after date of last dose, whichever is later
Description: AE that newly appears, increases in frequency, or worsens in severity following initiation of study drug and through the last study visit or up to 30
Groups:
- NEOD001 24 mg/kg: 24 mg/kg IV every 4 weeks for 12 months
- Placebo: 0.9% Saline IV every 4 weeks for 12 months
Arm/Group | NEOD001 24 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/66 | 6/63
Serious Adverse Events (participants affected / at risk) | 14/66 | 15/63
Other Adverse Events (participants affected / at risk) | 58/66 | 52/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=66) | Placebo (N=63)
Cardiac failure (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 4
Cellulitis (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 24 mg/kg (N=66) | Placebo (N=63)
Upper respiratory tract infection (Infections and infestations) | 6 | 8
Nasopharyngitis (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 6 | 3
Respiratory tract infection (Infections and infestations) | 5 | 2
Bronchitis (Infections and infestations) | 1 | 4
Fatigue (General disorders) | 14 | 14
Oedema peripheral (General disorders) | 7 | 8
Pyrexia (General disorders) | 4 | 4
Asthenia (General disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 11
Nausea (Gastrointestinal disorders) | 6 | 14
Constipation (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 6 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3
Headache (Nervous system disorders) | 9 | 6
Dizziness (Nervous system disorders) | 5 | 8
Hypoaesthesia (Nervous system disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Blood creatinine increased (Investigations) | 2 | 4
Hypocalcaemia (Investigations) | 3 | 4
Hyperuricaemia (Investigations) | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 6 | 11
Atrial fibrillation (Cardiac disorders) | 4 | 2
Hypertension (Vascular disorders) | 3 | 5
Hypotension (Vascular disorders) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 4
Haematuria (Renal and urinary disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI, institution and the sponsor have agreed that the PI and institution may publish or disclose study results from their site after the earlier of (a) publication of the complete multicenter study results or (b) 18 months after database lock for the multicenter study. The sponsor has at least 45 days to review a proposed publication and may request deletion of confidential information and up to 60 days additional delay to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2017-10-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT02632786/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT02632786/SAP_001.pdf